CLINICAL TRIAL: NCT04418284
Title: Evaluation of the Online Learning of Veterinary Anatomy During COVID-19 Pandemic
Brief Title: Online Learning of Veterinary Anatomy During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Mahdy, Principal Investigator, South Valley University
Other Study IDs: 2-2020
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: COVID-19; Anatomy; online learning
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Veterinary Medical students: Veterinary Medical students who are studying anatomy during COVID-19 pandemic lockdown
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — online survey

SUMMARY:
This study aims to analyze the online learning of veterinary anatomy during COVID-19 pandemic lockdown.

DETAILED DESCRIPTION:
Analysis of the online learning of veterinary anatomy during COVID-19 pandemic lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Veterinary Medical students who are studying anatomy online during the pandemic lockdown

Exclusion Criteria:

-

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Veterinary Medical students who are studying anatomy online during the pandemic lockdown
Sampling Method: Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Measure the students' interest in studying anatomy on-line. | 05/06/2020-05/07/2020
  An online questionnaire (Statement: I'm interested in studying anatomy on-line. Response: Strongly agree/ agree/ neutral/ disagree/ strongly disagree

SECONDARY OUTCOMES:
Assess the easiness of using technology during studying anatomy online | 05/06/2020-05/07/2020
  An online questionnaire (Statement: I'm comfortable with technological skills during online studying of anatomy. (Using Computers, surfing the internet, downloading files, etc.....) Response: Strongly agree/ agree/ neutral/ disagree/ strongly disagree)
Assess the student satisfaction regarding the provided study materials | 05/06/2020-05/07/2020
  1- An online questionnaire (Statement: The anatomy study materials provided to me by the lecturers were enough.
  Response: Strongly agree/ agree/ neutral/ disagree/ strongly disagree)

OTHER OUTCOMES:
Online learning as a substitution for face-to-face teaching | 05/06/2020-05/07/2020
  An online questionnaire (Statement: On-line learning of anatomy can replace face-to-face teaching. Response: Strongly agree/ agree/ neutral/ disagree/ strongly disagree
Measure the understanding of anatomy using on-line learning. | 05/06/2020-05/07/2020
  An online questionnaire (Statement:I can understand anatomy well using on-line learning.. Response: Strongly agree/ agree/ neutral/ disagree/ strongly disagree
Assess the average studying time of anatomy before and during the pandemic lockdown | 05/06/2020-05/07/2020
  1. A question: What is the average studying hours of anatomy before COVID-19 pandemic? Response: number of studying hours per week
  2. A question: What is the average studying hours of anatomy during COVID-19 pandemic? Response: number of studying hours per week
Assess the common problems during studying anatomy online | 05/06/2020-05/07/2020
  A question: What is the most common problem did you face during the online learning of anatomy?

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided